CLINICAL TRIAL: NCT03157687
Title: Detection of Luminal and Mucosa-associated Microbiome in Healthy Controls vs. Local and Systemic Inflammation Under Mixed Diet
Brief Title: Detection of Luminal and Mucosa-associated Microbiome in Healthy Controls vs. Local and Systemic Inflammation
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: MicrobiomStudy
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-01

CONDITIONS: Human Microbiome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: * Blood sampling for nutrition and inflammatory status
  * Stool sampling before preventive gastroscopy and colonoscopy
  * Questionnaires about general health, gastrointestinal symptoms and 3-day food record
  * Collection of biopsies in duodenum during gastroscopy
  * Collection of biopsies in terminal ileum, cecum, colon ascendens, sigma
- Inflammatory bowel disease (IBD): * Blood sampling for nutrition and inflammatory status
  * Stool sampling before indicated gastroscopy and colonoscopy
  * Questionnaires about general health, gastrointestinal symptoms and 3-day food record
  * Collection of biopsies in duodenum during gastroscopy
  * Collection of biopsies in terminal ileum, cecum, colon ascendens, sigma
- Liver transplantation recipient (LTX): * Blood sampling for nutrition and inflammatory status
  * Stool sampling before indicated gastroscopy and colonoscopy for evaluation of liver transplantation (LTX)
  * Questionnaires about general health, gastrointestinal symptoms and 3-day food record
  * Collection of biopsies in duodenum during gastroscopy
  * Collection of biopsies in terminal ileum, cecum, colon ascendens, sigma

SUMMARY:
This study should reveal differences in composition of luminal and mucosa-associated microbiome of the human gastrointestinal tract.Therefore bacterial species of different intestinal location sites (small intestine and colon) isolated of biopsies were compared to bacterial composition of stool samples. Additionally the bacterial composition of healthy persons, patients with inflammatory bowel disease and with liver disease (liver cirrhosis) will be compared to detect influence of local and systemic inflammation on microbiome.

DETAILED DESCRIPTION:
A dysbiosis of human gut microbiome is discussed in the pathogenesis of many disorders, also including gastrointestinal (e.g. inflammatory bowel disease, IBD) or liver diseases (e.g. liver cirrhosis) . A detailed analysis of intestinal bacterial patterns might reveal important findings for understanding disease pathogenesis. Thereby many studies only analysed the luminal microbiome of stool samples, whereas mucosa-associated bacteria have possibly a greater impact on human health and immune system .

To determine the differences of luminal and mucosa-associated bacteria, stool and mucosa samples (via biopsies) will be collected. Thereby biopsies are taken of different intestinal locations (small intestine and colon) to detect variations along intestinal tract. An additional comparison of bacterial patterns in patients with chronic, local (IBD) and systemic inflammation (with liver cirrhosis) or without intestinal inflammations (healthy controls) should reveal the influence of microbiome on or by inflammation processes.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with indication for cancer screening without gastrointestinal symptoms
* patients with inflammatory bowel disease (Crohn's disease and ulcerative colitis)
* patients with indication for evaluation of liver transplantation (LTX)

Exclusion Criteria:

* other gastrointestinal disease, e.g. celiac disease, gastrointestinal tumors
* antibiotic treatment within 6 weeks before gastroscopy / colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy controls patients with inflammatory bowel disease patients with liver disease (liver cirrhoses) and indication for LTX-evaluation
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
bacterial composition | 1 day
  detection of bacterial families in stool and mucosa samples

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No